CLINICAL TRIAL: NCT07252258
Title: Comparison of Frequency of Calcium Hydroxide Mixed With 0.2% Chlorhexidine Versus Saline as Intracanal Medicament in Periapical Periodontitis-A Randomized Controlled Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aqsa Afzal (Other)
Responsible Party: Sponsor-Investigator, Aqsa Afzal, FAyoub, College of Physicians and Surgeons Pakistan
Organization: College of Physicians and Surgeons Pakistan (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 118-ERB/023
Record Dates: First submitted 2025-11-19; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Periapical Periodontitis
MeSH Terms: conditions — Periapical Periodontitis | interventions — Calcium Hydroxide; Saline Solution; chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcium Hydroxide + Saline (Placebo Comparator): Participants in this arm will receive intracanal medicament consisting of calcium hydroxide mixed with normal saline after standard chemomechanical root canal preparation. Temporary restoration will be placed, and postoperative pain will be assessed at designated intervals
  Interventions: Drug: Calcium Hydroxide + Normal Saline
- Calcium Hydroxide + 0.2% Chlorhexidine (Experimental): Participants in this arm will receive intracanal medicament consisting of calcium hydroxide mixed with 0.2% chlorhexidine digluconate following standard root canal procedures. Temporary restoration will be placed, and postoperative pain will be evaluated.
  Interventions: Drug: Calcium Hydroxide + 0.2% Chlorhexidine Digluconate

INTERVENTIONS:
Drug: Calcium Hydroxide + Normal Saline — Calcium hydroxide powder mixed with sterile normal saline and placed inside the root canal as intracanal medicament.
  Arms: Calcium Hydroxide + Saline
Drug: Calcium Hydroxide + 0.2% Chlorhexidine Digluconate — Calcium hydroxide powder combined with 0.2% chlorhexidine solution and placed inside the root canal as intracanal medicament.
  Arms: Calcium Hydroxide + 0.2% Chlorhexidine

SUMMARY:
This randomized controlled trial aims to compare the effectiveness of calcium hydroxide mixed with 0.2% chlorhexidine digluconate versus calcium hydroxide mixed with saline as intracanal medicaments in reducing postoperative pain in patients with apical periodontitis. A total of 80 adult patients with anterior teeth diagnosed with apical periodontitis will be randomly assigned to two equal groups. After standard chemomechanical root canal preparation, Group A will receive calcium hydroxide with saline, while Group B will receive calcium hydroxide with 0.2% chlorhexidine. Postoperative pain will be assessed using a 10-point Visual Analogue Scale (VAS) at 12, 24, and 48 hours. The primary outcome is the frequency and severity of pain at 24 hours. Data will be analyzed using chi-square or Fisher's exact test, with a significance level of p < 0.05. The study aims to determine whether the addition of chlorhexidine improves the analgesic and antimicrobial effectiveness of calcium hydroxide during root canal treatment.

ELIGIBILITY:
Inclusion Criteria:

* • Patients age 18 or above 18 year old (to have complete apex formation)

  * Anterior teeth with apical periodontitis (simple root canal morphology)
  * Patients whose medical history does not include a history of certain illnesses, such as HIV, heart disease, or epilepsy (conditions that can affect a patient's rate of healing).

Exclusion Criteria:

* Patient allergic to chlorhexidine digluconate and Calcium hydroxide assessed by history.
* Tooth having necrotic pulp on radiographic examination and electric pulp tester.
* Multiple rooted teeth.
* Previously root canal treated tooth because of procedural errors and periapical infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
primary outcome measure | 24 hours after placement of intracanal medicament (pain also recorded at 12 and 48 hours, but final outcome measured at 24 hours).
  Postoperative pain will be assessed using a 10-point Visual Analogue Scale (VAS), where 0 = no pain, 1-3 = mild pain, 4-6 = moderate pain, and 7-10 = severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Saidu College of Dentistry Swat, Swāt, Khyber Pakhtunkhwa, Pakistan